CLINICAL TRIAL: NCT01130740
Title: Patient and Provider Interventions for Managing Osteoarthritis in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IIR 10-126
Record Dates: First submitted 2010-05-24; First posted 2010-05-26 (Estimated); Results first posted 2015-01-26 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2014-09

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; Exercise; Diet; Coping Skills; Education, Medical
MeSH Terms: conditions — Osteoarthritis; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (No Intervention): usual care
- Arm 2 (Experimental): Osteoarthritis Intervention - Primary care providers receive patient-specific osteoarthritis information and treatment recommendations approximately one week prior to the patient's first post-enrollment routine appointment with PCP; patients receive a 12-month intervention consisting of monthly phone calls focusing on exercise, weight management, and cognitive behavioral pain management.
  Interventions: Behavioral: Osteoarthritis Intervention

INTERVENTIONS:
Behavioral: Osteoarthritis Intervention — Primary care providers receive patient-specific osteoarthritis information and treatment recommendations two times (0 and 6 months); patients receive a 12-month intervention consisting of monthly phone calls focusing on exercise, weight management, and cognitive behavioral pain management.
  Arms: Arm 2

SUMMARY:
Osteoarthritis (OA) is one of the most common chronic conditions and a leading cause of disability among veterans. Many veterans with OA have significant pain and functional limitations, even though they receive some medical care for their OA. Efforts are needed to help veterans to improve OA-related outcomes. This study will examine a comprehensive approach to helping veterans manage their OA-related symptoms, in the context of a VA clinical setting. The study examines an intervention aimed at helping veterans with behaviors that are known to improve OA-related pain and function (such as exercise, weight management, and coping with pain), as well as helping providers to implement evidence-based recommendations for clinical care. The intervention is relatively low cost and easy to disseminate, with the patient component being telephone based. Therefore, if effective, this intervention could be implemented widely across the VA healthcare system.

DETAILED DESCRIPTION:
Evidence-based guidelines emphasize that adequate management of osteoarthritis (OA) requires a combination of both medical and behavioral modalities. However, many of the recommended guidelines are not regularly incorporated into clinical practice, and the recommended behavioral strategies (e.g. exercise and weight management) are not practiced by most patients. The objective of this study is examine the effectiveness of a combined intervention for patients (involving exercise, weight management, and cognitive behavioral pain management) and providers (involving provision of patient-specific recommendations for care, based on evidence-based guidelines) for improving OA-related outcomes in a real-world VA clinical setting. To our knowledge this is will be the first study to intervene at a both the patient and provider levels for managing OA.

This will be a randomized controlled trial of n=300 patients with symptomatic knee or hip OA, with equal assignment to 2 study arms: 1) Patient and Provider Intervention for OA and 2.) Usual Care Control. We will randomize 30 primary care providers at the Durham VAMC and affiliated community based outpatient clinics to either intervention or control groups. We will then enroll 10 patients from each provider (5 White, 5 Non-White). The patient component of the intervention will be a twelve-month program that includes the following elements: written educational materials (focused on exercise, weight management, and cognitive behavioral pain management), an exercise video tailored for patients with lower extremity OA, and telephone calls by a counselor to support behavior change. The provider component of the intervention will involve giving information on patients' OA symptoms and treatment, as well as patient-specific evidence-based recommendations for care. Providers will have access to this information, as well as facilitated referrals for patient-specific treatment recommendations (e.g. physical therapy, orthopedics), at the point of clinical care, via electronic medical records. The primary time point for outcome assessment will be at 12-months. We will also assess a limited set of outcomes via telephone at 6-months. The primary outcome will be the Western Ontario and McMasters Universities Osteoarthritis Index (WOMAC). Secondary outcomes will include objective physical function (Short Physical Performance Test) and depressive symptoms (PHQ-8). The main study analyses will compare outcomes between the intervention and control groups. We will also assess the cost-effectiveness of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* radiographic evidence of hip OA and / or radiographic of or meets clinical criteria for knee OA
* current joint symptoms
* BMI >=25
* physically inactive

Exclusion Criteria:

* Diagnosis of rheumatoid arthritis, fibromyalgia, or other systemic rheumatic disease
* Hospitalized for a stroke, myocardial infarction or coronary artery revascularization in the past 3 months
* Active diagnosis of psychosis or serious personality disorder
* On waiting list for / planning arthroplasty
* Severely impaired hearing or speech (patients must be able to respond to phone calls)
* Unable to speak English
* No access to a telephone
* Participating in another OA intervention or other lifestyle change study
* Dementia or other memory loss condition
* Current, uncontrolled substance abuse disorder
* Motor neuron diseases, Parkinson's Disease, multiple sclerosis
* Quadriplegic or paraplegic
* Serious / terminal illness as indicated by referral to hospice or palliative care
* Other self-reported health problem that would prohibit participation in the study
* Nursing home resident
* Other health conditions or personal issues judged by a study team member or primary care physician to make the patient inappropriate for the study
* Female participants: pregnant or planning to become pregnant
* Metastatic Cancer
* History of gout in knee or hip
* Total joint replacement (knee or hip) surgery, other knee or hip surgery, meniscus tear (verified by MRI), or ACL tear in the past 6 months
* Have not seen their VA-assigned primary health care provider for more than a year

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2011-08; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelli Dominick Allen, PhD, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

REFERENCES:
- [Result] Allen KD, Bosworth HB, Brock DS, Chapman JG, Chatterjee R, Coffman CJ, Datta SK, Dolor RJ, Jeffreys AS, Juntilla KA, Kruszewski J, Marbrey LE, McDuffie J, Oddone EZ, Sperber N, Sochacki MP, Stanwyck C, Strauss JL, Yancy WS Jr. Patient and provider interventions for managing osteoarthritis in primary care: protocols for two randomized controlled trials. BMC Musculoskelet Disord. 2012 Apr 24;13:60. doi: 10.1186/1471-2474-13-60. PMID 22530979
- [Result] Sperber N, Hall KS, Allen K, DeVellis BM, Lewis M, Callahan LF. The role of symptoms and self-efficacy in predicting physical activity change among older adults with arthritis. J Phys Act Health. 2014 Mar;11(3):528-35. doi: 10.1123/jpah.2012-0030. Epub 2013 Feb 8. PMID 23416927
- [Derived] Taylor SS, Hughes JM, Coffman CJ, Jeffreys AS, Ulmer CS, Oddone EZ, Bosworth HB, Yancy WS Jr, Allen KD. Prevalence of and characteristics associated with insomnia and obstructive sleep apnea among veterans with knee and hip osteoarthritis. BMC Musculoskelet Disord. 2018 Mar 9;19(1):79. doi: 10.1186/s12891-018-1993-y. PMID 29523117
- [Derived] Allen KD, Yancy WS Jr, Bosworth HB, Coffman CJ, Jeffreys AS, Datta SK, McDuffie J, Strauss JL, Oddone EZ. A Combined Patient and Provider Intervention for Management of Osteoarthritis in Veterans: A Randomized Clinical Trial. Ann Intern Med. 2016 Jan 19;164(2):73-83. doi: 10.7326/M15-0378. Epub 2015 Dec 22. PMID 26720751

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Primary care providers in the Durham VA Ambulatory Care Service and their patients were recrutied from this study. Recruitment began on August 4, 2011 and was completed on December 30, 2012.
Groups:
- Usual Care: Participants received no intervention durnig the study period but continued with any other usual care for osteoarthritis.
- Osteoarthritis Intervention: Osteoarthritis Intervention - Primary care providers receive patient-specific osteoarthritis information and treatment recommendations approximately one week prior to the patient's first post-enrollment routine appointment with PCP; patients receive a 12-month intervention consisting of monthly phone calls focusing on exercise, weight management, and cognitive behavioral pain management.
  Osteoarthritis Intervention: Primary care providers receive patient-specific osteoarthritis information and treatment recommendations two times (0 and 6 months); patients receive a 12-month intervention consisting of monthly phone calls focusing on exercise, weight management, and cognitive behavioral pain management.
Period: Overall Study
Arm/Group | Usual Care | Osteoarthritis Intervention
Started | 149 | 151
Completed | 137 | 136
Not Completed | 12 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Osteoarthritis Intervention | Total
Number analyzed (Participants) | 149 | 151 | 300
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (9.0) | 60.4 (9.4) | 61.1 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 20 | 28
  Male | 141 | 131 | 272
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 65 | 69 | 134
  White | 73 | 67 | 140
  More than one race | 8 | 12 | 20
  Unknown or Not Reported | 2 | 1 | 3
Western Ontario and McMasters Universities Osteoarthritis Index (WOMAC) [Mean (Standard Deviation); unit: units on a scale] — The WOMAC includes 24 items, each measured on a Likert Scale of 0-4, with a range of 0-96 and higher scores indicating worse symptoms. There are 3 subscales that make up the total scale:pain (5 items), stiffness (2 items) and function (17 items).
  units on a scale | 47.8 (17.4) | 48.9 (17.6) | 48.4 (17.5)
Short Performance Physical Test [Mean (Standard Deviation); unit: units on a scale] — Objective functional tests, including an 8-foot timed walk, chair stands, and a series of three balance tests.
  units on a scale | 8.1 (2.48) | 8.0 (2.63) | 8.0 (2.6)
Patient Health Questionnaire 8 (PHQ-8) [Mean (Standard Deviation); unit: units on a scale] — 8-item validated, self-report measure of depressive symptoms.
  units on a scale | 6.4 (5.13) | 7.2 (5.57) | 6.8 (5.36)

OUTCOME MEASURES:

1. Primary Outcome: Western Ontario and McMasters Universities Osteoarthritis Index (WOMAC)
Description: Self-report measure of lower extremity pain (5 items), stiffness (2 items), and function (17 items) in the past two weeks. All items are rated on a 5-point Likert scale ranging from "none" (0) to "severe / extreme" (4), for a total of range of 0-96. Higher scores indicate worse symptoms and poorer function. The Mixed Models Analysis described below utilizes a common baseline mean rather than means for the individual arms. This common baseline mean is presented here, and the raw baseline measures per group are presented in the baseline information section.
Time Frame: 12-months
Population: All enrolled participants were analyzed, on an intent to treat basis. One enrolled participants in the Usual Care grouped changed clinical care to an enrolled OA Intervention provider after randomization, so that participant was analyzed with the OA intervention group.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Usual Care | Osteoarthritis Intervention
Number analyzed (Participants) | 149 | 151
units on a scale
  Common Baseline | 48.4 (1.09) | 48.4 (1.09)
  6-Month | 43.5 (1.45) | 41.2 (1.47)
  12-Month | 48.5 (1.38) | 44.4 (1.39)
Statistical Analysis 1: Comparison: Usual Care vs Osteoarthritis Intervention; This is a comparison of 6-month outcomes between the two study groups. (Primary comparison is for 12 months.); Test type: Superiority or Other; p = 0.158, Mixed Models Analysis
Statistical Analysis 2: Comparison: Usual Care vs Osteoarthritis Intervention; This is the 12-month comparison between the 2 study groups, which is the primary study analysis; Test type: Superiority or Other; p = 0.008, Mixed Models Analysis

2. Secondary Outcome: Short Physical Performance Test Protocol
Description: This is a series of 5 tests covering the domains of balance (3 tests), gait speed (8 foot walk) and time to rise from a chair and return to the seated position five times. The total score ranges from 0 (worst performance) to 12 (best performance).
  The Mixed Models Analysis described below utilizes a common baseline mean rather than means for the individual arms. This common baseline mean is presented here, and the raw baseline measures per group are presented in the baseline information section.
Time Frame: 12-months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Usual Care | Osteoarthritis Intervention
Number analyzed (Participants) | 149 | 151
units on a scale
  Common Baseline | 8.01 (0.149) | 8.01 (0.149)
  12 Months | 7.53 (0.233) | 7.86 (0.237)
Statistical Analysis 1: Comparison: Usual Care vs Osteoarthritis Intervention; This is the between-group 12-month comparison; Test type: Superiority or Other; p = 0.274, Mixed Models Analysis

3. Secondary Outcome: PHQ-8
Description: This is an 8-item self-report scale, all items are rated on a score of 0-3, for a total range of 0-24. Higher scores indicate more depressive symptoms. The Mixed Models Analysis described below utilizes a common baseline mean rather than means for the individual arms. This common baseline mean is presented here, and the raw baseline measures per group are presented in the baseline information section.
Time Frame: 12-months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Usual Care | Osteoarthritis Intervention
Number analyzed (Participants) | 149 | 151
units on a scale
  Common Baseline | 6.83 (0.31) | 6.83 (0.31)
  12 Months | 6.83 (0.39) | 6.21 (0.39)
Statistical Analysis 1: Comparison: Usual Care vs Osteoarthritis Intervention; Test type: Superiority or Other; p = 0.177, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: For each participant, the collection period was 1 year: baseline to 12-month follow-up.
Arm/Group | Usual Care | Osteoarthritis Intervention
Serious Adverse Events (participants affected / at risk) | 18/149 | 25/151
Other Adverse Events (participants affected / at risk) | 9/149 | 44/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Usual Care (N=149) | Osteoarthritis Intervention (N=151)
Hospitalization (Blood and lymphatic system disorders) | 5 | 6 — The intervention group had more regular contact with the study team than the usual care group. In some cases this resulted in higher rates of non-systematic reporting of serious but not study related adverse events for the intervention group.
Hospitalization (Gastrointestinal disorders) | 0 | 6 — The intervention group had more regular contact with the study team than the usual care group. In some cases this resulted in higher rates of non-systematic reporting of serious but not study related adverse events for the intervention group.
Hospitalization (Hepatobiliary disorders) | 0 | 1 — The intervention group had more regular contact with the study team than the usual care group. In some cases this resulted in higher rates of non-systematic reporting of serious but not study related adverse events for the intervention group.
Hospitalization (Infections and infestations) | 0 | 2 — The intervention group had more regular contact with the study team than the usual care group. In some cases this resulted in higher rates of non-systematic reporting of serious but not study related adverse events for the intervention group.
Hospitalization (Injury, poisoning and procedural complications) | 0 | 10 — The intervention group had more regular contact with the study team than the usual care group. In some cases this resulted in higher rates of non-systematic reporting of serious but not study related adverse events for the intervention group.
Hospitalization (Musculoskeletal and connective tissue disorders) | 0 | 1 — The intervention group had more regular contact with the study team than the usual care group. In some cases this resulted in higher rates of non-systematic reporting of serious but not study related adverse events for the intervention group.
Outpatient Surgery (Musculoskeletal and connective tissue disorders) | 2 | 0 — The intervention group had more regular contact with the study team than the usual care group. In some cases this resulted in higher rates of non-systematic reporting of serious but not study related adverse events for the intervention group.
Emergency Room Visit (Musculoskeletal and connective tissue disorders) | 1 | 0 — The intervention group had more regular contact with the study team than the usual care group. In some cases this resulted in higher rates of non-systematic reporting of serious but not study related adverse events for the intervention group.
Hospitalization (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 — The intervention group had more regular contact with the study team than the usual care group. In some cases this resulted in higher rates of non-systematic reporting of serious but not study related adverse events for the intervention group.
Hospitalization (Nervous system disorders) | 1 | 0 — The intervention group had more regular contact with the study team than the usual care group. In some cases this resulted in higher rates of non-systematic reporting of serious but not study related adverse events for the intervention group.
Hospitalization (Psychiatric disorders) | 1 | 0 — The intervention group had more regular contact with the study team than the usual care group. In some cases this resulted in higher rates of non-systematic reporting of serious but not study related adverse events for the intervention group.
Hospitalization (Renal and urinary disorders) | 0 | 1 — The intervention group had more regular contact with the study team than the usual care group. In some cases this resulted in higher rates of non-systematic reporting of serious but not study related adverse events for the intervention group.
Hospitalization (Respiratory, thoracic and mediastinal disorders) | 0 | 3 — The intervention group had more regular contact with the study team than the usual care group. In some cases this resulted in higher rates of non-systematic reporting of serious but not study related adverse events for the intervention group.
Hospitalization (Surgical and medical procedures) | 5 | 11 — The intervention group had more regular contact with the study team than the usual care group. In some cases this resulted in higher rates of non-systematic reporting of serious but not study related adverse events for the intervention group.
Outpatient Surgery (Surgical and medical procedures) | 6 | 7 — The intervention group had more regular contact with the study team than the usual care group. In some cases this resulted in higher rates of non-systematic reporting of serious but not study related adverse events for the intervention group.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Usual Care (N=149) | Osteoarthritis Intervention (N=151)
Emergency Room Visit (Blood and lymphatic system disorders) | 0 | 2 — The intervention group had more regular contact with the study team than the usual care group. In some cases this resulted in higher rates of non-systematic reporting of non-serious and not study related adverse events for the intervention group.
Emergency Room Visit (Cardiac disorders) | 2 | 3 — The intervention group had more regular contact with the study team than the usual care group. In some cases this resulted in higher rates of non-systematic reporting of non-serious and not study related adverse events for the intervention group.
Emergency Room Visit (Ear and labyrinth disorders) | 1 | 1 — The intervention group had more regular contact with the study team than the usual care group. In some cases this resulted in higher rates of non-systematic reporting of non-serious and not study related adverse events for the intervention group.
Emergency Room Visit (Endocrine disorders) | 3 | 3 — The intervention group had more regular contact with the study team than the usual care group. In some cases this resulted in higher rates of non-systematic reporting of non-serious and not study related adverse events for the intervention group.
Emergency Room Visit (Eye disorders) | 0 | 1 — The intervention group had more regular contact with the study team than the usual care group. In some cases this resulted in higher rates of non-systematic reporting of non-serious and not study related adverse events for the intervention group.
Emergency Room Visit (Gastrointestinal disorders) | 2 | 5 — The intervention group had more regular contact with the study team than the usual care group. In some cases this resulted in higher rates of non-systematic reporting of non-serious and not study related adverse events for the intervention group.
Emergency Room Visit (General disorders) | 2 | 4 — The intervention group had more regular contact with the study team than the usual care group. In some cases this resulted in higher rates of non-systematic reporting of non-serious and not study related adverse events for the intervention group.
Emergency Room Visit (Infections and infestations) | 1 | 4 — The intervention group had more regular contact with the study team than the usual care group. In some cases this resulted in higher rates of non-systematic reporting of non-serious and not study related adverse events for the intervention group.
Emergency Room Visit (Injury, poisoning and procedural complications) | 1 | 3 — The intervention group had more regular contact with the study team than the usual care group. In some cases this resulted in higher rates of non-systematic reporting of non-serious and not study related adverse events for the intervention group.
Emergency Room Visit (Musculoskeletal and connective tissue disorders) | 4 | 22 — The intervention group had more regular contact with the study team than the usual care group. In some cases this resulted in higher rates of non-systematic reporting of non-serious and not study related adverse events for the intervention group.
Emergency Room Visit (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 — The intervention group had more regular contact with the study team than the usual care group. In some cases this resulted in higher rates of non-systematic reporting of non-serious and not study related adverse events for the intervention group.
Emergency Room Visit (Nervous system disorders) | 0 | 6 — The intervention group had more regular contact with the study team than the usual care group. In some cases this resulted in higher rates of non-systematic reporting of non-serious and not study related adverse events for the intervention group.
Emergency Room Visit (Psychiatric disorders) | 1 | 2 — The intervention group had more regular contact with the study team than the usual care group. In some cases this resulted in higher rates of non-systematic reporting of non-serious and not study related adverse events for the intervention group.
Emergency Room Visit (Renal and urinary disorders) | 0 | 8 — The intervention group had more regular contact with the study team than the usual care group. In some cases this resulted in higher rates of non-systematic reporting of non-serious and not study related adverse events for the intervention group.
Emergency Room Visit (Reproductive system and breast disorders) | 0 | 1 — The intervention group had more regular contact with the study team than the usual care group. In some cases this resulted in higher rates of non-systematic reporting of non-serious and not study related adverse events for the intervention group.
Emergency Room Visit (Respiratory, thoracic and mediastinal disorders) | 3 | 11 — The intervention group had more regular contact with the study team than the usual care group. In some cases this resulted in higher rates of non-systematic reporting of non-serious and not study related adverse events for the intervention group.
Emergency Room Visit (Skin and subcutaneous tissue disorders) | 1 | 2 — The intervention group had more regular contact with the study team than the usual care group. In some cases this resulted in higher rates of non-systematic reporting of non-serious and not study related adverse events for the intervention group.
Emergency Room Visit (Surgical and medical procedures) | 1 | 0 — The intervention group had more regular contact with the study team than the usual care group. In some cases this resulted in higher rates of non-systematic reporting of non-serious and not study related adverse events for the intervention group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes